CLINICAL TRIAL: NCT00924924
Title: Act Healthy! A Controlled Trial of Worksite Health Promotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 1141037
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: health promotion; prevention; worksite wellness; behavior change; healthy volunteers
MeSH Terms: interventions — Self-Management; Health Promotion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Act Healthy! (Experimental): Immediate treatment group of six-weeks of classes in self-management training for healthy behaviors
  Interventions: Behavioral: Act Healthy!
- Delayed treatment control (Active Comparator): Delayed self-management training group - begins following completion of the experimental group training
  Interventions: Behavioral: Act Healthy!; Behavioral: Delayed treatment control

INTERVENTIONS:
Behavioral: Act Healthy! — Six-week class of 50 minute sessions of self-management training for health behaviors
  Other Names: self-management; health promotion; worksite wellness; behavior change
Behavioral: Delayed treatment control — Delayed self-management training group - begins following completion of the experimental group training
  Arms: Delayed treatment control

SUMMARY:
The purpose of this project is to determine if a worksite wellness intervention using a theoretically-based self-management model increases confidence for carrying out healthy behaviors and improves health practices of participating employees. The research questions are: 1) does the intervention produce between group differences in behavior self-efficacy and actual health behaviors, 2) are self-efficacy and performance of health behaviors related, and 3) do changes in self-efficacy result in changes in behavior.

DETAILED DESCRIPTION:
The purpose of this project is to see if a six-week education program called Act Healthy! led by trained volunteers from the UM T.E. Atkins Wellness Program is able to help people who take the classes improve their confidence in their ability to choose good health behaviors and carry out new behaviors. The project will use the Stanford University Self-management education model and train volunteers to be teachers. People who work on the MU campus will be recruited to take a 50-minute class once a week for six weeks. Class members will complete questionnaires before and after the class and again three months later that ask about their health behaviors and confidence to perform health behaviors. This information will be analyzed to determine if the classes were effective in helping people act in healthier ways.

ELIGIBILITY:
Inclusion Criteria:

* full-time employee of the University of Missouri

Exclusion Criteria:

* inability to read and speak in English

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Self-report of health behaviors | pre-, post intervention; 3-month follow up

SECONDARY OUTCOMES:
self-efficacy for health behaviors | pre- and post-intervention; 3-month follow up
Stages of change scale | pre- and post-intervention; 3-month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Marian A Minor, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No